CLINICAL TRIAL: NCT00001426
Title: A Multi-Institutional Phase II Study of Cyclophosphamide, Paclitaxel, Cisplatin With G-CSF for Patients With Newly Diagnosed Advanced Stage Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 950055; 95-C-0055; NCT00019045 (obsolete NCT alias)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2013-11-07

CONDITIONS: Ovarian Neoplasm
Keywords: Ovarian Cancer; Initial Therapy; Paclitaxel; Cisplatin; Cyclophosphamide
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Cyclophosphamide; Paclitaxel; Cisplatin; Granulocyte Colony-Stimulating Factor

INTERVENTIONS:
Drug: Cyclophosphamide
Drug: Paclitaxel
Drug: Cisplatin
Drug: G-CSF

SUMMARY:
A supra-additive cytotoxic effect was seen when CAI and paclitaxel were given to human ovarian cancer cells sequentially in tissue culture. We have demonstrated that CAI given for 8 days followed by paclitaxel is reasonably well tolerated and that paclitaxel administration causes a dose-dependent increase in CAI plasma concentration. CAI is a cytostatic drug and continuous exposure is needed. This study will evaluate the combination of continuously administered CAI with three-weekly paclitaxel.

DETAILED DESCRIPTION:
A supra-additive cytotoxic effect was seen when CAI and paclitaxel were given to human ovarian cancer cells sequentially in tissue culture. We have demonstrated that CAI given for 8 days followed by paclitaxel is reasonably well tolerated and that paclitaxel administration causes a dose-dependent increase in CAI plasma concentration. CAI is a cytostatic drug and continuous exposure is needed. This study will evaluate the combination of continuously administered CAI with three-weekly paclitaxel.

ELIGIBILITY:
* INCLUSION CRITERIA:

All patients must have biopsy proven, newly diagnosed epithelial ovarian cancer, primary epithelial fallopian tube cancer, or peritoneal surface carcinoma. Histopathologic diagnosis must be confirmed in the pathology department of the treating institution prior to initiation of therapy. Diagnosis will be confirmed in the Laboratory of Pathology, National Cancer Institute. This confirmation is not necessary prior to entering the patient onto protocol.

Patients must have FIGO stage III or IV disease and will undergo attempted surgical debulking prior to the initiation of chemotherapy.

Patients must be able to begin therapy within 6 weeks of staging laparotomy and should have an indwelling venous access device placed. A double lumen catheter is preferred.

Performance status of less than or equal to ECOG 2.

Patients must be able to give written informed consent and express a willingness to meet all of the expected requirements of the protocol.

All patients must be registered by calling the Orkand Corporation at 301-402-1732 between the hours of 8:30 AM and 5:00 PM EST; Eligibility criteria will be queried.

EXCLUSION CRITERIA:

Evidence CNS involvement (patients with normal clinical exam will not require a head CT scan or MRI).

History of myocardial infarction or unstable dysrhythmia within 1 month of study entry.

Creatinine clearance of less than 60 cc/min, ANC less than 1000/cm3, platelet count less than 1000,000/cm3.

History of active GI bleeding within the last 30 days.

Prior therapy other than surgery for this malignancy.

Abnormal PT, PTT, and bilirubin. SGOT greater than or equal to 3 times the upper limit of normal.

Previous history of invasive malignancy.

Patients with ureteral obstruction must have this corrected prior to starting therapy.

Patients with germ cell, mixed Muellerian and borderline histologies are specifically excluded.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 1995-02-03; Primary Completion 2007-10-15 (Actual); Study Completion 2013-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elise C Kohn, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kohn EC, Sarosy GA, Davis P, Christian M, Link CE, Ognibene FP, Sindelar WF, Jacob J, Steinberg SM, Premkumar A, Reed E. A phase I/II study of dose-intense paclitaxel with cisplatin and cyclophosphamide as initial therapy of poor-prognosis advanced-stage epithelial ovarian cancer. Gynecol Oncol. 1996 Aug;62(2):181-91. doi: 10.1006/gyno.1996.0213. PMID 8751547
- [Background] Reed E, Kohn EC, Sarosy G, Dabholkar M, Davis P, Jacob J, Maher M. Paclitaxel, cisplatin, and cyclophosphamide in human ovarian cancer: molecular rationale and early clinical results. Semin Oncol. 1995 Jun;22(3 Suppl 6):90-6. PMID 7541159
- [Background] Link CJ Jr, Sarosy GA, Kohn EC, Christian MC, Davis P, Adamo DO, Reed E. Cutaneous manifestations of Taxol therapy. Invest New Drugs. 1995;13(3):261-3. doi: 10.1007/BF00873811. PMID 8729957